CLINICAL TRIAL: NCT04585594
Title: Mi Propio Camino (Finding My Own Way): Personalized Approaches to Improve Blood Pressure Control
Brief Title: Mi Propio Camino Intervention RCT for Blood Pressure Medication Adherence
Acronym: MPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John Thomas Billimek, Faculty, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20174025; 1R01HL142964 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Medication Adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mi Propio Camino (MPC; My Own Way) (Experimental): Participants will complete the MPC intervention alongside usual care for hypertension
  Interventions: Behavioral: Mi Propio Camino (MPC)
- Habilidades para Controlar la Presion (HCP; Skills for Blood Pressure Control) (Active Comparator): Participants will complete the HCP intervention alongside usual care for hypertension.
  Interventions: Behavioral: Habilidades para Controlar la Presion (HCP; Skills for Blood Pressure Control)

INTERVENTIONS:
Behavioral: Mi Propio Camino (MPC) — The Mi Propio Camino (MPC) intervention will be comprised of four sessions. Session 1 will encompass: the facts about high blood pressure (BP), understanding blood pressure readings, provide an overview of changes one can make to manage their BP, introduce MPC personal experience monitoring, and usage the mHealth kit. Subsequently, sessions 2-4 will emphasize the benefits of personal experience monitoring through 1) personal insight (finding what works for them) and 2) empowerment to work with their providers. Session 2 will reinforce this by introducing: synergy between medication and lifestyle, principles of heart-healthy eating and physical activity. Session 3 will incorporate discussion of negative beliefs about medication and patient directed lifestyle learning-rotating stations. Lastly, session 4 will introduce the continuation of personal experience monitoring on their own through the use of behavioral strategies for adherence and provider communication strategies.
  Other Names: MPC
  Arms: Mi Propio Camino (MPC; My Own Way)
Behavioral: Habilidades para Controlar la Presion (HCP; Skills for Blood Pressure Control) — The HCP intervention will be comprised of four sessions and introduce seven lifestyle strategies (LS) subdivided per these sessions. Session 1 will encompass the facts about high blood pressure (BP), understanding blood pressure readings, provide an overview of changes one can make to manage their BP, present specific health threats from high BP, and incorporate LS1: taking control of your medication. Subsequently, sessions 2-4 will reinforce the benefits of taking medications through presenting 1) reduced risk for complications and 2) strategies to remember to take medications. Session 2 will present LS2: eating a well-balanced, low-salt diet and LS3: enjoying regular physical activity. Session 3 will follow with introducing LS4: maintaining a healthy weight and LS5: shaking the salt habit while eating out. Session 4 will present LS6: managing stress and LS7: working together with their doctor followed by a review of strategies they can continue on their own.
  Other Names: HCP
  Arms: Habilidades para Controlar la Presion (HCP; Skills for Blood Pressure Control)

SUMMARY:
The purpose of this study is to compare the effect of two educational interventions on adherence to blood pressure medications among adults with uncontrolled hypertension.

DETAILED DESCRIPTION:
The study is a randomized controlled trial (RCT) consisting of a 4-session educational intervention (completed over the course of 4-8 weeks) and a 6-month follow-up period for adherence monitoring. Participants will be allocated to one of two educational intervention groups following a block randomization schedule, stratified on the hypothesized mediator variable of medication-related beliefs (high versus low scores on the BMQ Necessity-Concerns subscore) to ensure the groups are balanced on this variable. Primary endpoint is medication adherence at 6 month follow-up, defined as the proportion of days that the prescribed number of doses was taken by the patient during a 30-day period, measured by a pill bottle cap monitor (medication events monitoring device [MEMS]).

ELIGIBILITY:
Inclusion criteria are: (1) age 18 years or greater, (2) uncontrolled hypertension (BP above 140/90 mmHg), (3) Hispanic ethnicity, (4) Spanish or English-speaking, (5) at least one office visit at the study clinic in prior 12 months.

Exclusion criteria: Persons with stage 4 or 5 chronic kidney disease (CKD) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Medication Adherence (Objective) | 6 months post-intervention
  Medication adherence is assessed at 6-month follow-up with Medication Event Monitoring System (MEMS) pill bottle cap monitors (MWV/WestRock), an objective, gold-standard measure for pill-taking behavior. MEMS caps can be affixed to a medicine bottle to record each time the bottle is opened, indicating when the patient took the medication. Daily adherence is defined as the proportion of days that the prescribed number of doses was taken by the patient during a 30-day period.

SECONDARY OUTCOMES:
Blood Pressure | Blood pressure will be collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  This outcome measure will be recorded following the American Heart Association (AHA) and American College of Cardiology (ACC) guidelines for proper methods and accurate blood pressure (BP) measurement. Accurate BP measurements are subdivided into pre and post-steps. Before measuring of BP, patients are to be prepared for proper technique including: having the patient sit quietly with their feet on the floor, back supported and relaxed for 5 minutes, supporting arm used for measurement on a desk and ensuring it is positioned at heart level. Subsequently, the middle of the BP cuff should be positioned on the patient's upper arm ensuring that the correct cuff size is used based on the cuff size criteria from AHA. As our patients are already taking medication that might affect BP, timing of measurements should be standardized to the patient's medication intake.
Medication Adherence (Subjective) | Collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  Subjective medication adherence assessed with a validated Spanish version of the Morisky Medication Adherence Scale (8-item MMAS), coded dichotomously (low vs. high adherence) using published cutoffs
Reasons for Nonadherence | Collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  Reasons for medication nonadherence will be assessed with the Safran Medication Adherence questionnaire, coded dichotomously for nonadherence related to beliefs, nonadherence related to cost, and unintentional nonadherence
Medication-related beliefs (Specific) | Collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  Medication-related beliefs will be assessed as the Specific Necessity-Concerns scale for the Beliefs about Medicines Questionnaire (BMQ).
Medication-related information | Collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  Knowledge of medication-related information will be assessed with a questionnaire adapted from the Medication Knowledge Questionnaire (MKQ)
Medication-related Behavioral Skills | Collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  Knowledge of Medication-related Behavioral Skills will be assessed withthe PROMIS Self-Efficacy for Managing Chronic Conditions Manage Medications/Treatment scale
Activation of behavioral strategies | Collected for analysis at baseline, upon completion of intervention period and upon completion of outcome assessment period at 1-month and 6-month follow up.
  Activation of behavioral strategies measured with the Medication Adherence Strategies Inventory (ASI)60, an inventory of 7 common strategies for adherence.

CONTACTS AND LOCATIONS:
Overall Officials: John Billimek, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Health Policy Research Institute, Irvine, California, United States